CLINICAL TRIAL: NCT02863081
Title: Helping Older Persons Emerge Stronger (HOPES) After Intensive Care Unit Admission
Brief Title: Helping Older Persons Emerge Stronger
Acronym: HOPES
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Select Medical (Unknown)
Responsible Party: Principal Investigator, Michele Balas, Associate Professor College of Nursing, Ohio State University
Other Study IDs: 2016H0001
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Delirium; Ventilators; Pain; Agitation; Anxiety
MeSH Terms: conditions — Delirium; Pain; Psychomotor Agitation; Anxiety Disorders | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthcare providers: All healthcare providers working in the participating LTACH will be asked to complete 2 surveys and invited to participate in focus group meetings
  Interventions: Other: Survey; Other: interview
- Patients: 81 LTACH patients will be enrolled over the course of a 9 month period. Each patient and their LAR will be interviewed at the time of LTACH admission to garner information about their pre hospitalization physical, functional, and cognitive health status. Each day enrolled patients will undergo daily symptom assessments and medical record reviews. At the time of LTACH discharge all enrolled patients will be interviewed again to garner information about their discharge physical, functional, and cognitive health status.
  Interventions: Other: interview

INTERVENTIONS:
Other: Survey — Administered to healthcare providers
  Other Names: Focus group interviews
  Groups: Healthcare providers
Other: interview — Administered to patients and LAR (i.e., interviews)
  Other Names: symptom assessment; Medical record review

SUMMARY:
Select Specialty, a national network of more than 100 LTACHs across the United States, has expressed the desire to adopt the ABCDEF bundle as a "standard of care" for its patients. As part of this initiative, Select first plans to conduct an ABCDEF bundle quality improvement project in one of its local hospitals. The overall purpose of this before-after study is to study prospectively the process and effects of implementing the ABCDEF bundle into the everyday care of patients requiring prolonged mechanical ventilation in the LTACH setting.

DETAILED DESCRIPTION:
The 300,000 chronically critically ill patients each year who require prolonged mechanical ventilation (PMV)1,2 represent an ever-growing, extremely vulnerable, proportion of intensive care unit (ICU) survivors.3 The increasing number of these patients is an important factor in the expanded use of long-term acute care hospitals (LTACHs), centers that specialize in mechanical ventilation weaning and rehabilitation. The 412 LTACHs currently operated in the United States admit more than 130,000 patients annually and account for more than $5 billion in Medicare expenditures each year.4,5 Unfortunately, LTACH stays for patients requiring PMV are typically complicated and associated with a number of poor outcomes including very high one-year mortality rates (44-77%),6,7 severe and enduring brain dysfunction (i.e., coma and/or delirium), life-altering functional decline, substantial pain and suffering, caregiver burden and diminished quality of life.6-11 While returning home is often an important goal for patients and their families,3 this is a rare outcome in this population.11 Rather, patients requiring PMV often experience multiple transitions in care in the year following their original hospital admission (median of 4), which results in further costs and persistent, profound disability.9 Despite these disheartening findings, to date there is very limited scientific evidence available to help clinicians care for the chronically critically ill, particularly those requiring PMV in LTACHs.

Chronically critically ill patients are generally older, sicker and have more comorbidities than their acutely ill counterparts.12 Importantly, they also suffer from much greater symptom burden, with up to 90% of patients experiencing at least one distressing symptom during the course of their illness (e.g., pain, dyspnea, weakness).13 While these symptoms are often thought of as unfortunate and inevitable consequences of critical illness,14 evidence suggests that the inappropriate management of these symptoms may actually be causal to the poor outcomes experienced by this group.15 For example, the results of numerous, well-designed, clinical trials conducted in the traditional ICU setting by our team and others suggest regular pain, agitation, and delirium assessment, prevention and treatment, coupled with strategies that decrease patients' exposure to sedative medications, support early mobilization, promote evidence-based mechanical ventilation discontinuation approaches, and actively engage and empower family members in patient care can positively affect important patient-centered outcomes (e.g., improved survival and physical/cognitive ability).16-26 One unifying method of implementing these evidence based interventions into everyday practice is consistent and reliable use of the ABCDEF bundle (i.e., Assess, prevent, and manage pain, Both Spontaneous Awakening Trials (SATs) & Spontaneous Breathing Trials (SBTs), Choice of analgesia and sedation, Delirium assess, prevent, and manage, Early mobility and exercise, and Family engagement and empowerment).27 Congruent with the Society of Critical Care Medicine's Clinical Practice Guidelines for the Management of Pain, Agitation, and Delirium and endorsed by a number of patient safety and quality organizations including the Institute for Healthcare Improvement and the Gordon and Betty Moore Foundation, the ABCDEF bundle is being actively implemented in ICUs throughout the world. The strength of evidence supporting the ABCDEF bundle, coupled with this strong implementation momentum, has prompted interest in the LTACH in applying the bundle into the everyday care of chronically critically ill patients who require mechanical ventilation.

Select Specialty, a national network of more than 100 LTACHs across the United States, has expressed the desire to adopt the ABCDEF bundle as a "standard of care" for its patients. As part of this initiative, Select first plans to conduct an ABCDEF bundle quality improvement project in one of its local hospitals. The overall purpose of this before-after study is to study prospectively the process and effects of implementing the ABCDEF bundle into the everyday care of patients requiring prolonged mechanical ventilation in the LTACH setting. Specifically the study's aims are to:

Aim 1: Identify facilitators and barriers to successful ABCDEF bundle implementation in the LTACH setting.

Aim 2: Compare the symptom experience (e.g., pain, agitation, anxiety, fatigue, shortness of breath, restlessness, sadness, hunger, fear, thirst, confusion sedative medication exposure) of patients receiving usual LTACH care (during months 1-4.5) to those treated with the ABCDEF bundle (during months 4.5-9).

Aim 3. Evaluate the impact ABCDEF bundle implementation has on safety (i.e., new pneumonias, device self-removal) and patient-centered outcomes (i.e., delirium/coma free days, weaning duration, tracheostomy removal , mortality, depression, post-traumatic stress disorder, functional and cognitive ability, discharge disposition, opioid and benzodiazepine withdrawal rates, and quality of life) of patients receiving usual LTACH care (during months 1-4.5) to those treated with the ABCDEF bundle (during months 4.5-9).

To complete these aims the investigators will administer an on-line survey and conduct focus group interviews with LTACH staff before and after the ABCDEF bundle is implemented into everyday care. Over the course of a nine month period, the investigators will also consent and enroll 81 patients who require mechanical ventilation at the time of LTACH admission. These patients will undergo daily, in-person symptom assessment using valid and reliable screening tools. Finally, medical record reviews and brief patient interviews will be conducted to obtain data on our outcomes of interest.

ELIGIBILITY:
Aim 1:

Inclusion • All full and part-time Registered Nurses, attending physicians, respiratory therapists, pharmacists, and physical/occupational/speech therapists who regularly care for patients requiring prolonged mechanical ventilation in the LTACH setting

Exclusion

• None

Aims 2 and 3:

Inclusion

* >18 years old
* Admitted to the LTACH with a tracheostomy
* Require mechanical ventilation > 8 hours a day upon LTACH admission
* English speaking

Exclusion Criteria:

* Severe neurologic deficits defined as coma (i.e., Richmond Agitation Sedation Score < -4 or -5 due to stroke, intracranial hemorrhage, cranial trauma, malignancy, anoxic brain injury, or cerebral edema)
* Inability to obtain informed consent from the patient's legally authorized representative (LAR) within 72 hours of meeting all inclusion criteria
* Chronic ventilator dependence that is deemed "not weanable" by admitting LTACH physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Healthcare providers working in a LTACH
  2. Chronically critically ill patients requiring mechanical ventilation at the time of LTACH admission
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Facilitators/Barriers to successful ABCDEF bundle implementation in the LTACH setting | 9 months
  Achieved through surveys and focus groups of LTACH providers
Pain | 9 months
  As measured by numeric rating scale of behavioral pain sclae
All cause mortality | 9 months

SECONDARY OUTCOMES:
Level of Arousal | 9 months
  As measured by Richmond Agitation and Sedation Scale (RASS)
Delirium | 9 months
  As measured by Confusion Assessment Method ICU (CAM-ICU)
Anxiety Anxiety | 9 months
  As measured by Visual Analog Scale
Other Symptoms | 9 month
  As measured by Patient Symptom Survey
Opioid Withdrawal | 9 months
  As measured by Clinical Opiate WIthdrawl Scale
Benzodiazepine Withdrawal | 9 months
  As measured by Clinical Institute Withdrawal Assessment Scale-Benzodiazepines
Delirium/Coma free days | 9 months
  As measured by CAM ICU and RASS
Weaning duration | 9 months
New Pneumonia | 9 months
Device self-removal | 9 months
Tracheostomy removal | 90 months
Depression | 90 months
  As measured by Hospital Anxiety and Depression Scale
Post Traumatic Stress Disorder | 9 months
  As measured by Impact of Event Scale
Functional ability | 9 months
  As measured by Functional Status Score ICU, KATZ ADL, LAWTON IADL
Cognitive ability | 9 months
  As measure by Mini Mental State Exam
Quality of Life | 9 months
  As measured by SF 36

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No